CLINICAL TRIAL: NCT06095726
Title: Comparative Effect of Peppermint Inhalation and Swedish Massage on Chemotherapy Induced-Nausea and Vomiting in Children With Leukemia.
Brief Title: Peppermint Inhalation Versus Swedish Massage on Chemotherapy Induced-Nausea and Vomiting in Children With Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CINV
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Leukemia
Keywords: leukemia; Swedish Massage; Peppermint Inhalation; Nausea; Vomiting; Chemotherapy; Children
MeSH Terms: conditions — Leukemia; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Children with leukemia received routine nursing and hospital care for management of chemotherapy induced nausea and vomiting (antiemetic medications only).
- Peppermint Inhalation Group (Experimental): Children with leukemia received the inhalation of essential oil of peppermint 2% in addition to routine nursing and hospital care for management of chemotherapy induced nausea and vomiting.
  Interventions: Behavioral: Peppermint Inhalation
- Swedish Massage Group: (Experimental): Children with leukemia received the Swedish massage therapy in addition to routine nursing and hospital care for management of chemotherapy induced nausea and vomiting.
  Interventions: Behavioral: Swedish Massage

INTERVENTIONS:
Behavioral: Peppermint Inhalation — The researcher applied two drops (0,2ml) of 2% essential oil of peppermint on a piece of cotton. Then, each child was instructed to take three breaths of the essence that had been put on a piece of cotton before starting chemotherapy session with three minutes. In addition, the piece of cotton with peppermint essence was kept at bed side table to use by child as needed throughout the chemotherapy session. Inhalation of peppermint essence was applied for three consecutive chemotherapy sessions.
  Arms: Peppermint Inhalation Group
Behavioral: Swedish Massage — Children were received Swedish massage therapy for twenty minutes prior to chemotherapy session in a private and special room with effleurage, petrissage, friction, and tapotement and vibration movements for three consecutive chemotherapy sessions. The researcher applied facilitating olive oil in hands and pre warmed before applying massage. The massage technique was applied in prone position with mild to moderate pressure with guidance by the child's feedback and tolerance by using non-scented olive oil. Children's privacy was considered.
  Arms: Swedish Massage Group:

SUMMARY:
Clinical trials was used to compare the effect of peppermint inhalation and Swedish massage on chemotherapy induced-nausea and vomiting in children with leukemia. the main research hypotheses are:

* Children with leukemia who receive peppermint inhalation exhibit less chemotherapy induced- nausea and vomiting than those who don't receive.
* Children with leukemia who receive Swedish massage exhibit less chemotherapy induced-nausea and vomiting than those who don't receive.
* Children with leukemia who receive Swedish massage exhibit less chemotherapy induced- nausea and vomiting than those who receive peppermint inhalation. children divided into three groups of study ( control group, peppermint inhalation group and Swedish massage group) to identify its effect on chemotherapy induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Received first chemotherapy session
* Intact skin in the massage

Exclusion Criteria:

* Chronic and acute disorders such as respiratory, cardiovascular diseases...etc.
* Allergy from any essential oils.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Experience of anticipatory nausea | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  Yes/No
Worst of anticipatory nausea | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  No/Mild/Moderate/severe/intolerable
Duration of anticipatory nausea | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  /Minutes
Frequency of anticipatory nausea | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  once/twice/ three times and more
Experience of anticipatory vomiting | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  Yes/No
Worst of anticipatory vomiting | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  No/Mild/Moderate/severe/intolerable
Amount of anticipatory vomiting | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  Small/ Moderate/ Large
Frequency of anticipatory vomiting | assessed immediately before chemotherapy administration for three consecutive chemotherapy sessions
  once/ twice/ three times and more.
Experience of acute nausea . | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  Yes/no.
Worst of acute nausea . | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  No/Mild/Moderate/severe/intolerable
Duration of acute nausea . | Frst 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  /hours.
Frequency of acute nausea . | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  once/ twice/ three times and more.
Experience of acute vomiting. | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  Yes/No.
Worst of acute vomiting. | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  No/Mild/Moderate/severe/intolerable
Amount of acute vomiting. | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  Small/ Moderate/ large
Frequency of acute vomiting. | First 24 hours after first chemotherapy administration of study. Assessed within the first 24 hours after second chemotherapy administration of study. Assessed within the first 24 hours after third chemotherapy administration of study.
  once/ twice/ three times and more.
Experience of delayed nausea. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  Yes/ No.
Worst of delayed nausea. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  No/Mild/Moderate/severe/intolerable
Duration of delayed nausea. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  /hours.
Frequency of delayed nausea. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  once/ twice/ three times and more.
Experience of delayed vomiting. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  Yes/ No.
Worst of delayed vomiting. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  No/Mild/Moderate/severe/intolerable
Amount of delayed vomiting. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  Small/ Moderate/ large
Frequency of delayed vomiting. | On second and third days after first chemotherapy administration.On second and third days after second chemotherapy administration. On second and third days after third chemotherapy administration.
  once/ twice/ three times and more.

OTHER OUTCOMES:
Child's age | Before data collection
  years
Gender | Before data collection
  male/female
Residence | Before data collection
  rural/urban
Level of education | Before data collection
  kinder garden/primary
Onset of the disease | Before data collection
  months
Type of leukemia | Before data collection
  Acute Lymphoblastic Leukemia / Acute Myeloid Leukemia/ Chronic Lymphocytic Leukemia / Chronic Myeloid Leukemia
Prescribed chemotherapy medications | Before data collection
  Methotrexate / cytarabine
Antiemetics prescribed medications | Before data collection
  Ondansetron

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Arafa Badr, Alexandria, Egypt

REFERENCES:
- [Background] Sowmiya Rajendran, Ruthrani Princely J, Kanchana S, Celina D., Effectiveness of Swedish Massage on the Level of Chemotherapy Induced Nausea and Vomiting (CINV) Among Children with Cancer at a Selected Hospital in North India, ICCRJNR, Jul - Dec 2016, 1(2): 20-38.
- [Background] Evans A, Malvar J, Garretson C, Pedroja Kolovos E, Baron Nelson M. The Use of Aromatherapy to Reduce Chemotherapy-Induced Nausea in Children With Cancer: A Randomized, Double-Blind, Placebo-Controlled Trial. J Pediatr Oncol Nurs. 2018 Nov/Dec;35(6):392-398. doi: 10.1177/1043454218782133. Epub 2018 Jun 27. PMID 29947285
- [Background] El-SayedYousef, Y., Zaki, N. A., AsmaaAbd-Alasis, Abdel-RazikSayed, H., & Elsayed, F. (2018). Effect of Therapeutic Massage on nausea and vomitingamong Children with Leukemia following Chemotherapy.
- [Result] Ahmad, M. (2016). Tool Development to Assess Nausea and Vomiting Among Patients Receiving Chemotherapy. International Journal of Cancer and Oncology, 3(1), 1-5. https://doi.org/10.15436/2377-0902.16.031